CLINICAL TRIAL: NCT04460755
Title: Tooth Whitening Evaluation With Cytotoxic and Genotoxic Effect of Commercial Whitening Toothpastes on Oral Mucosal Cells
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Zagreb (Other)
Responsible Party: Principal Investigator, Nada Zorica Vladislavic, Tooth Whitening Evaluation With Cytotoxic and Genotoxic Effect of Commercial Whitening Toothpastes on Oral Mucosal Cells, University of Zagreb
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 05-PA-30-9/2018.; 2181-198-03-04-17-0063 (Other Grant/Funding Number: School of Medicine, University of Split)
Record Dates: First submitted 2020-06-27; First posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Teeth Whitening
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The study is randomized, prospective clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Control group (Active Comparator): A group of participants that will be using toothpaste without tooth whitening ingredients.
  Interventions: Other: Control group
- Whitening toothpaste 1 (Experimental): A group of participants that will be using urea peroxide whitening toothpastes.
  Interventions: Other: Whitening toothpaste 1
- Whitening toothpaste 2 (Experimental): A group of participants that will be using hydrogen peroxide whitening toothpastes.
  Interventions: Other: Whitening toothpaste 2
- Whitening toothpaste 3 (Experimental): A group of participants that will be using whitening toothpastes that contain abrasive ingredients.
  Interventions: Other: Whitening toothpaste 3
- Whitening toothpaste 4 (Experimental): A group of participants that will be using whitening toothpastes that contain enzymes as whitening ingredients.
  Interventions: Other: Whitening toothpaste 4
- Whitening toothpaste 5 (Experimental): A group of participants that will be using toothpastes that contain an activated charcoal.
  Interventions: Other: Whitening toothpaste 5

INTERVENTIONS:
Other: Control group — A sample of cells from the buccal mucosa area will be taken with cytological sampling brush and will be fixed on on a microscopy slide and stained with a Feulgen fast green solution. The samples will be analyzed by electron microscopy. Tooth color will be measured, verified and evaluated with a Vita Easyshade V digital spectrophotometer in initial phase, after one month of usage, after two months of usage and one month after the end of usage.
  Before using any of the whitening toothpaste under test, every participant will use non whitening toothpaste for one month, twice a day.
  Satisfaction and impression with treatment will be recorded with the questionnaires provided for this study.
  Arms: Control group
Other: Whitening toothpaste 1 — A sample of cells from the buccal mucosa area will be taken with cytological sampling brush and will be fixed on on a microscopy slide and stained with a Feulgen fast green solution. The samples will be analyzed by electron microscopy. Tooth color will be measured, verified and evaluated with a Vita Easyshade V digital spectrophotometer in initial phase, after one month of usage, after two months of usage and one month after the end of usage.
  Before using any of the whitening toothpaste under test, every participant will use non whitening toothpaste for one month, twice a day.
  Satisfaction and impression with treatment will be recorded with the questionnaires provided for this study.
  Arms: Whitening toothpaste 1
Other: Whitening toothpaste 2 — A sample of cells from the buccal mucosa area will be taken with cytological sampling brush and will be fixed on on a microscopy slide and stained with a Feulgen fast green solution. The samples will be analyzed by electron microscopy. Tooth color will be measured, verified and evaluated with a Vita Easyshade V digital spectrophotometer in initial phase, after one month of usage, after two months of usage and one month after the end of usage.
  Before using any of the whitening toothpaste under test, every participant will use non whitening toothpaste for one month, twice a day.
  Satisfaction and impression with treatment will be recorded with the questionnaires provided for this study.
  Arms: Whitening toothpaste 2
Other: Whitening toothpaste 3 — A sample of cells from the buccal mucosa area will be taken with cytological sampling brush and will be fixed on on a microscopy slide and stained with a Feulgen fast green solution. The samples will be analyzed by electron microscopy. Tooth color will be measured, verified and evaluated with a Vita Easyshade V digital spectrophotometer in initial phase, after one month of usage, after two months of usage and one month after the end of usage.
  Before using any of the whitening toothpaste under test, every participant will use non whitening toothpaste for one month, twice a day.
  Satisfaction and impression with treatment will be recorded with the questionnaires provided for this study.
  Arms: Whitening toothpaste 3
Other: Whitening toothpaste 4 — A sample of cells from the buccal mucosa area will be taken with cytological sampling brush and will be fixed on on a microscopy slide and stained with a Feulgen fast green solution. The samples will be analyzed by electron microscopy. Tooth color will be measured, verified and evaluated with a Vita Easyshade V digital spectrophotometer in initial phase, after one month of usage, after two months of usage and one month after the end of usage.
  Before using any of the whitening toothpaste under test, every participant will use non whitening toothpaste for one month, twice a day.
  Satisfaction and impression with treatment will be recorded with the questionnaires provided for this study.
  Arms: Whitening toothpaste 4
Other: Whitening toothpaste 5 — A sample of cells from the buccal mucosa area will be taken with cytological sampling brush and will be fixed on on a microscopy slide and stained with a Feulgen fast green solution. The samples will be analyzed by electron microscopy. Tooth color will be measured, verified and evaluated with a Vita Easyshade V digital spectrophotometer in initial phase, after one month of usage, after two months of usage and one month after the end of usage.
  Before using any of the whitening toothpaste under test, every participant will use non whitening toothpaste for one month, twice a day.
  Satisfaction and impression with treatment will be recorded with the questionnaires provided for this study.
  Arms: Whitening toothpaste 5

SUMMARY:
Bleaching discolored vital teeth is one of the most popular aesthetic treatment in dentistry in the last decade. Teeth whitening can be performed by professionals/dentists in the dental office ("in-office") and by the patients themselves at home (over-the-counter). A generally available method for teeth whitening is to use toothpastes which contain whitening ingredients. This method presents commercial option to remove discolorations on the enamel surface of vital teeth. There are many commercially available dentifrices that contain whitening agents, such as abrasives, chemical or optical agents. It has been noticed that whitening agents added in toothpastes can provide whitening effect visible to human eye that can objectively be evaluated by using sprectrophotometers. The results of teeth whitening can also be obtained subjectively by observation and comparison to tooth shade guide. Also, these products must be used with caution as they may cause some negative effects, such as dentinal hypersensitivity, irritations, peeling/exfoliation, dry mouth, rougher teeth and cytotoxic and genotoxic effect on oral mucosa cells. Studies that have already been conducted with whitening agents are based on abrasives, peroxides, optical agents and activated charcoal.

The main objective in this study is to investigate the effectiveness of different brands of toothpastes with whitening effect and their performance (effect) on oral mucosa cells. As a measure of genotoxicity and cytotoxicity in cells, the number of micronuclei and other morphological changes of the nucleus are determined (micronucleus assay). Other specific objectives are to investigate the patient satisfaction with the characteristic of treatment such as final tooth color, color stability, length of treatment, comfort during treatment and overall participant satisfaction.

DETAILED DESCRIPTION:
Sample description and study design for this research was performed at the School of the Medicine, University of Split, Croatia.

Respondents are the students and employees of the School of the Medicine University of Split, Croatia. They will be divided in groups where different types of whitening toothpaste will be used. One group will use control non-whitening toothpaste. All respondents will use the same toothbrush during the research. Before using whitening toothpastes, all participants will use the same non-whitening toothpaste for one month. All participants will sign informed consent for participation in the research. Their participation will be voluntary. Respondents will be able to refuse to participate in the research without any consequences.

This study is approved by Ethic Committee of the School of Dental Medicine, Zagreb, Croatia (09.2018.) and Ethic Committee of the School of the Medicine University of Split, Croatia (12.2017). The study is randomized, prospective clinical trial.

The participants will be randomly selected for the whitening toothpaste groups and for the control non-whitening group. A sample of cells from the buccal mucosa area will be taken from each patient prior using the toothpastes under test, 30 and 60 days after the beginning and 30 days after using the toothpastes under test. Color assessment will be performed four times using the Vita Easyshade digital spectrophotometer: T0- before treatment (initial); T1- 30 days after the beginning; T2- 60 days after the beginning and T3- 90 days after the beginning of the study (i.e. 30 days after completing the treatment). The color reading will be performed in the middle third of the labial surface of the tooth, in the same environment and with the same light conditions. The measurement will be performed on all vital six anterior maxillary teeth, free of caries and restorations. Participant's satisfaction with the treatment and the toothpaste used will be assessed using the prepared questionnaires.

Participants will use toothpastes under test for two months. Toothpaste will be applied twice a day, in the morning and in the evening, for three minutes for 1g (app. 2 cm). During the experiment, the examinees will not use any toothpaste other than the one under test. Participants will use no other agents for oral hygiene.

ELIGIBILITY:
Inclusion Criteria:

* age of 18 and older
* non smokers
* good oral and general health
* excellent oral hygiene
* vital six anterior maxillary teeth free of caries or restorations
* tooth shade A2 or darker
* no cervical lesions or prosthodontic treatments
* no periodontal disease

Exclusion Criteria:

* pregnant women
* breastfeeding women
* individuals with discolored teeth (tetracycline stain, fluorosis)
* tooth sensitivity
* history of allergy to any dental hygiene product
* individuals who had previously undergone any tooth whitening treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Color assessment before the treatment (T0) | 0 days
  The following measurements were will be recorded: L*,a*, b* values for all teeth as well as the tooth shade. The color was will be established by CIELAB color space. ΔE is will be calculated using the following formula: ΔE=√(〖(ΔL*)〗^2+〖(Δa*)〗^2+〖(Δb*)〗^2 ). The color changes between the evaluation times in each tested group and between groups were will be analysed using the ΔE, ΔL*, Δa* and Δb*values. To calculate the difference in tooth shade according to the Vita Classical scale, the recorded values were will be ordered in scores from 1 to 16 in a luminosity sequence.
Color change after 30 days of treatment (T1) | 30 days
  The following measurements were will be recorded: L*,a*, b* values for all teeth as well as the tooth shade. The color was will be established by CIELAB color space. ΔE is will be calculated using the following formula: ΔE=√(〖(ΔL*)〗^2+〖(Δa*)〗^2+〖(Δb*)〗^2 ). The color changes between the evaluation times in each tested group and between groups were will be analysed using the ΔE, ΔL*, Δa* and Δb*values. To calculate the difference in tooth shade according to the Vita Classical scale, the recorded values were will be ordered in scores from 1 to 16 in a luminosity sequence.
Color change after 60 days of treatment (T2) | 60 days
  The following measurements were will be recorded: L*,a*, b* values for all teeth as well as the tooth shade. The color was will be established by CIELAB color space. ΔE is will be calculated using the following formula: ΔE=√(〖(ΔL*)〗^2+〖(Δa*)〗^2+〖(Δb*)〗^2 ). The color changes between the evaluation times in each tested group and between groups were will be analysed using the ΔE, ΔL*, Δa* and Δb*values. To calculate the difference in tooth shade according to the Vita Classical scale, the recorded values were will be ordered in scores from 1 to 16 in a luminosity sequence.
Color change 30 days after the treatment (90 days from the beginning of treatment) (T3) | 90 days
  The following measurements were will be recorded: L*,a*, b* values for all teeth as well as the tooth shade. The color was will be established by CIELAB color space. ΔE is will be calculated using the following formula: ΔE=√(〖(ΔL*)〗^2+〖(Δa*)〗^2+〖(Δb*)〗^2 ). The color changes between the evaluation times in each tested group and between groups were will be analysed using the ΔE, ΔL*, Δa* and Δb*values. To calculate the difference in tooth shade according to the Vita Classical scale, the recorded values were will be ordered in scores from 1 to 16 in a luminosity sequence.
Assessment of biocompatibility before the treatment (T0) | 0 days
  Assessment of biocompatibility through cytotoxicity and genotoxicity parameters of commercially available toothpastes with whitening effect will be performed using micronucleus assay.
Assessment of biocompatibility after 30 days of treatment (T1) | 30 days
  Assessment of biocompatibility through cytotoxicity and genotoxicity parameters of commercially available toothpastes with whitening effect will be performed using micronucleus assay.
Assessment of biocompatibility after 60 days of treatment (T2) | 60 days
  Assessment of biocompatibility through cytotoxicity and genotoxicity parameters of commercially available toothpastes with whitening effect will be performed using micronucleus assay.
Assessment of biocompatibility 30 days after the treatment (90 days from the beginning of treatment) (T3) | 90 days
  Assessment of biocompatibility through cytotoxicity and genotoxicity parameters of commercially available toothpastes with whitening effect will be performed using micronucleus assay.

SECONDARY OUTCOMES:
Assessment of participant's satisfaction with treatment and used toothpaste after 60 days of treatment | 60 days
  Assessment of participant's satisfaction with treatment and used toothpaste will be performed by prepared questionnaire for the study. Respondents will complete a questionnaire of eating and living habits, too
Assessment of participant's satisfaction with treatment of used toothpaste 30 days after the treatment (90 days from the beginning of treatment) | 90 days
  Assessment of participant's satisfaction with treatment and used toothpaste will be performed by prepared questionnaire for the study.

CONTACTS AND LOCATIONS:
Locations (1):
- School of the Medicine, University of Split, Split, Croatia

REFERENCES:
- [Background] Joiner A. Whitening toothpastes: a review of the literature. J Dent. 2010;38 Suppl 2:e17-24. doi: 10.1016/j.jdent.2010.05.017. Epub 2010 May 24. PMID 20562012
- [Background] Epple M, Meyer F, Enax J. A Critical Review of Modern Concepts for Teeth Whitening. Dent J (Basel). 2019 Aug 1;7(3):79. doi: 10.3390/dj7030079. PMID 31374877
- [Background] van Loveren C, Duckworth RM. Anti-calculus and whitening toothpastes. Monogr Oral Sci. 2013;23:61-74. doi: 10.1159/000350698. Epub 2013 Jun 28. PMID 23817060
- [Background] Lippert F. An introduction to toothpaste - its purpose, history and ingredients. Monogr Oral Sci. 2013;23:1-14. doi: 10.1159/000350456. Epub 2013 Jun 28. PMID 23817056
- [Background] Pickles MJ, Evans M, Philpotts CJ, Joiner A, Lynch RJ, Noel N, Laucello M. In vitro efficacy of a whitening toothpaste containing calcium carbonate and perlite. Int Dent J. 2005;55(3 Suppl 1):197-202. doi: 10.1111/j.1875-595x.2005.tb00060.x. PMID 16004254
- [Background] Collins LZ, Naeeni M, Schafer F, Brignoli C, Schiavi A, Roberts J, Colgan P. The effect of a calcium carbonate/perlite toothpaste on the removal of extrinsic tooth stain in two weeks. Int Dent J. 2005;55(3 Suppl 1):179-82. doi: 10.1111/j.1875-595x.2005.tb00056.x. PMID 16004250
- [Background] Kalliath C, Mukunda A, Pynadath M, Venugopal V, Prethweeraj J. Comparison between the effect of commercially available chemical teeth whitening paste and teeth whitening paste containing ingredients of herbal origin on human enamel. Ayu. 2018 Apr-Jun;39(2):113-117. doi: 10.4103/ayu.AYU_82_18. PMID 30783367
- [Background] Patil PA, Ankola AV, Hebbal MI, Patil AC. Comparison of effectiveness of abrasive and enzymatic action of whitening toothpastes in removal of extrinsic stains - a clinical trial. Int J Dent Hyg. 2015 Feb;13(1):25-9. doi: 10.1111/idh.12090. Epub 2014 Jul 21. PMID 25046241
- [Background] Kalyana P, Shashidhar A, Meghashyam B, Sreevidya KR, Sweta S. Stain removal efficacy of a novel dentifrice containing papain and Bromelain extracts--an in vitro study. Int J Dent Hyg. 2011 Aug;9(3):229-33. doi: 10.1111/j.1601-5037.2010.00473.x. Epub 2010 Jul 1. PMID 21356017
- [Background] Hara AT, Turssi CP. Baking soda as an abrasive in toothpastes: Mechanism of action and safety and effectiveness considerations. J Am Dent Assoc. 2017 Nov;148(11S):S27-S33. doi: 10.1016/j.adaj.2017.09.007. PMID 29056187
- [Background] Ghassemi A, Hooper W, Vorwerk L, Domke T, DeSciscio P, Nathoo S. Effectiveness of a new dentifrice with baking soda and peroxide in removing extrinsic stain and whitening teeth. J Clin Dent. 2012;23(3):86-91. PMID 23210419
- [Background] Vaz VTP, Jubilato DP, Oliveira MRM, Bortolatto JF, Floros MC, Dantas AAR, Oliveira Junior OB. Whitening toothpaste containing activated charcoal, blue covarine, hydrogen peroxide or microbeads: which one is the most effective? J Appl Oral Sci. 2019 Jan 14;27:e20180051. doi: 10.1590/1678-7757-2018-0051. PMID 30673027
- [Background] Franco MC, Uehara J, Meroni BM, Zuttion GS, Cenci MS. The Effect of a Charcoal-based Powder for Enamel Dental Bleaching. Oper Dent. 2020 Nov 1;45(6):618-623. doi: 10.2341/19-122-L. PMID 32243248
- [Background] Joiner A, Luo W. Tooth colour and whiteness: A review. J Dent. 2017 Dec;67S:S3-S10. doi: 10.1016/j.jdent.2017.09.006. Epub 2017 Sep 18. PMID 28928097
- [Background] Korifi R, Le Dreau Y, Antinelli JF, Valls R, Dupuy N. CIEL*a*b* color space predictive models for colorimetry devices--analysis of perfume quality. Talanta. 2013 Jan 30;104:58-66. doi: 10.1016/j.talanta.2012.11.026. Epub 2012 Nov 23. PMID 23597889
- [Background] Martin J, Rivas V, Vildosola P, Moncada L, Oliveira Junior OB, Saad JR, Fernandez E, Moncada G. Personality Style in Patients Looking for Tooth Bleaching and Its Correlation with Treatment Satisfaction. Braz Dent J. 2016 Jan-Feb;27(1):60-5. doi: 10.1590/0103-6440201600127. PMID 27007348
- [Background] Paravina RD, Perez MM, Ghinea R. Acceptability and perceptibility thresholds in dentistry: A comprehensive review of clinical and research applications. J Esthet Restor Dent. 2019 Mar;31(2):103-112. doi: 10.1111/jerd.12465. Epub 2019 Mar 20. PMID 30891913
- [Background] Parameswaran V, Anilkumar S, Lylajam S, Rajesh C, Narayan V. Comparison of accuracies of an intraoral spectrophotometer and conventional visual method for shade matching using two shade guide systems. J Indian Prosthodont Soc. 2016 Oct-Dec;16(4):352-358. doi: 10.4103/0972-4052.176537. PMID 27746599
- [Background] Paravina RD, Powers JM, Fay RM. Dental color standards: shade tab arrangement. J Esthet Restor Dent. 2001;13(4):254-63. doi: 10.1111/j.1708-8240.2001.tb00271.x. PMID 11572509
- [Background] Chu SJ, Trushkowsky RD, Paravina RD. Dental color matching instruments and systems. Review of clinical and research aspects. J Dent. 2010;38 Suppl 2:e2-16. doi: 10.1016/j.jdent.2010.07.001. Epub 2010 Aug 1. PMID 20621154
- [Background] Paul S, Peter A, Pietrobon N, Hammerle CH. Visual and spectrophotometric shade analysis of human teeth. J Dent Res. 2002 Aug;81(8):578-82. doi: 10.1177/154405910208100815. PMID 12147751
- [Background] Camargo SE, Joias RP, Santana-Melo GF, Ferreira LT, El Achkar VN, Rode Sde M. Conventional and whitening toothpastes: cytotoxicity, genotoxicity and effect on the enamel surface. Am J Dent. 2014 Dec;27(6):307-11. PMID 25707084
- [Background] Holland N, Bolognesi C, Kirsch-Volders M, Bonassi S, Zeiger E, Knasmueller S, Fenech M. The micronucleus assay in human buccal cells as a tool for biomonitoring DNA damage: the HUMN project perspective on current status and knowledge gaps. Mutat Res. 2008 Jul-Aug;659(1-2):93-108. doi: 10.1016/j.mrrev.2008.03.007. Epub 2008 Apr 11. PMID 18514568
- [Background] Thomas P, Fenech M. Buccal micronucleus cytome assay. Methods Mol Biol. 2011;682:235-48. doi: 10.1007/978-1-60327-409-8_17. PMID 21057932
- [Background] Torres-Bugarin O, Zavala-Cerna MG, Nava A, Flores-Garcia A, Ramos-Ibarra ML. Potential uses, limitations, and basic procedures of micronuclei and nuclear abnormalities in buccal cells. Dis Markers. 2014;2014:956835. doi: 10.1155/2014/956835. Epub 2014 Feb 4. PMID 24778463
- [Background] Bolognesi C, Knasmueller S, Nersesyan A, Thomas P, Fenech M. The HUMNxl scoring criteria for different cell types and nuclear anomalies in the buccal micronucleus cytome assay - an update and expanded photogallery. Mutat Res. 2013 Oct-Dec;753(2):100-113. doi: 10.1016/j.mrrev.2013.07.002. Epub 2013 Aug 11. PMID 23942275
- [Background] Tolbert PE, Shy CM, Allen JW. Micronuclei and other nuclear anomalies in buccal smears: methods development. Mutat Res. 1992 Feb;271(1):69-77. doi: 10.1016/0165-1161(92)90033-i. PMID 1371831
- [Background] Tadin A, Gavic L, Zeravica A, Ugrin K, Galic N, Zeljezic D. Assessment of cytotoxic and genotoxic effects of conventional and whitening kinds of toothpaste on oral mucosa cells. Acta Odontol Scand. 2018 Jan;76(1):64-70. doi: 10.1080/00016357.2017.1384567. Epub 2017 Sep 29. PMID 28959909
- [Background] Tadin A, Gavic L, Govic T, Galic N, Zorica Vladislavic N, Zeljezic D. In vivo evaluation of fluoride and sodium lauryl sulphate in toothpaste on buccal epithelial cells toxicity. Acta Odontol Scand. 2019 Jul;77(5):386-393. doi: 10.1080/00016357.2019.1577988. Epub 2019 Feb 20. PMID 30784350
- [Background] Tadin A, Galic N, Mladinic M, Marovic D, Kovacic I, Zeljezic D. Genotoxicity in gingival cells of patients undergoing tooth restoration with two different dental composite materials. Clin Oral Investig. 2014 Jan;18(1):87-96. doi: 10.1007/s00784-013-0933-3. Epub 2013 Feb 5. PMID 23385426
- [Background] Akarslan ZZ, Sadik B, Erten H, Karabulut E. Dental esthetic satisfaction, received and desired dental treatments for improvement of esthetics. Indian J Dent Res. 2009 Apr-Jun;20(2):195-200. doi: 10.4103/0970-9290.52902. PMID 19553722
- [Background] Sabherwal RS, Gonzalez J, Naini FB. Assessing the influence of skin color and tooth shade value on perceived smile attractiveness. J Am Dent Assoc. 2009 Jun;140(6):696-705. doi: 10.14219/jada.archive.2009.0256. PMID 19491166
- [Background] Kershaw S, Newton JT, Williams DM. The influence of tooth colour on the perceptions of personal characteristics among female dental patients: comparisons of unmodified, decayed and 'whitened' teeth. Br Dent J. 2008 Mar 8;204(5):E9; discussion 256-7. doi: 10.1038/bdj.2008.134. Epub 2008 Feb 15. PMID 18297050
- [Background] Angel P, Bersezio C, Estay J, Werner A, Retamal H, Araya C, Martin J, Fernandez E. Color stability, psychosocial impact, and effect on self-perception of esthetics of tooth whitening using low-concentration (6%) hydrogen peroxide. Quintessence Int. 2018;49(7):557-566. doi: 10.3290/j.qi.a40468. PMID 29786702
- [Derived] Vladislavic NZ, Vladislavic J, Franic I, Tadin A. Cytotoxicity and genotoxicity of whitening toothpastes in buccal mucosal cells: a randomized controlled trial. Clin Oral Investig. 2023 Oct;27(10):6245-6259. doi: 10.1007/s00784-023-05241-6. Epub 2023 Sep 14. PMID 37704916
- [Derived] Vladislavic NZ, Tadin A, Gavic L, Jerkovic D, Franic I, Verzak Z. In vivo evaluation of whitening toothpaste efficiency and patient treatment satisfaction: a randomized controlled trial. Clin Oral Investig. 2022 Jan;26(1):739-750. doi: 10.1007/s00784-021-04052-x. Epub 2021 Jul 10. PMID 34245356